CLINICAL TRIAL: NCT05154786
Title: The Effects of Early Mobilization and Endurance Training for Patients With Prolonged Mechanical Ventilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Chi-Wen Lin, Physical Therapist, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC108-28
Record Dates: First submitted 2021-10-29; First posted 2021-12-13 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Mechanical Ventilation Complication
Keywords: Mechanical Ventilators; Weaning; Exercise therapy
MeSH Terms: interventions — Early Ambulation; Endurance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Mobilization and endurance training (Experimental): Early Mobilization and endurance training for prolonged mechanical ventilator
  Interventions: Other: Early Mobilization and endurance training
- Usual care (Active Comparator): Weaning protocols, bed exercise, and early mobilization.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Early Mobilization and endurance training — The early mobilization and endurance training will be conducted with grading exercise level. In the course of endurance training. After achieving patient's active participation in sitting on the bed, the goal will be to train for at least 20 min. If this is accomplished, exercise level and training period increased until a maximum of 7 on modified RPE. If these are well-tolerated and no contraindications as per medical prescription exist, the treatment will be further advanced to mobilizing participants to the bedside. After being able to sit for at least 10 min on the side of the bed, regardless of whether support is needed, participants will be moved into a chair with an individually adapted transfer according to the individual's resources.While sitting, functional tasks and activities of daily living will be performed and gradually increased to standing and walking exercises.
  Arms: Early Mobilization and endurance training
Other: Usual Care — The weaning protocols, bed exercise, positioning, respiratory therapy, and early mobilization.
  Arms: Usual care

SUMMARY:
The primary hypothesis is that prolonged mechanically ventilated adults who participate in an early mobilization and endurance exercise training protocol, have an improved pulmonary outcome and functional capacity and more functionally independent at hospital discharge compared to patients receiving the usual physiotherapy care. Further, the investigators expect improvements in weaning rate from mechanical ventilator, less time on mechanical ventilation, a shorter length of stay in the respiratory care center and the hospital, and a higher quality of life at 6 months after hospital discharge compared to patients receiving usual care. The investigators will conduct a prospective, single-center, allocation concealed and assessor-blinded randomised controlled trial with superiority design and 6-month follow-up. The study is being conducted in the interdisciplinary respiratory care center of Taichung Tzu Chi Hospital, Taiwan. To be eligible to participate in the study patients must be aged 18 to 75, be expected to stay on mechanical ventilator for at least 21 days, which reflects a prolonged stay at mechanical ventilator. Standard care (control group) Participants randomised to the control group will receive usual physiotherapy and respiratory care center standard care, which includes weaning protocols and bed exercise program based on previous publications. In this procedure, physiotherapy and mobilization will start after medical prescription. Treatments are based on the therapist's assessment and are accordingly individually tailored. Sessions will usually take place once daily from Monday to Friday. The participants randomised to the experimental group will receive a standardised exercise program involving early mobilization and endurance training.

The endurance training will be conducted with grading exercise level. In the course of endurance training, The participants will be prompted verbally for at least 10 min. The aim during all mobilizations will be to involve the participants as actively as possible to promote independence.

DETAILED DESCRIPTION:
The primary hypothesis is that prolonged mechanically ventilated adults who participate in an early mobilization and endurance exercise training protocol, have an improved pulmonary outcome and functional capacity and are, therefore, more functionally independent at hospital discharge compared to patients receiving the usual physiotherapy care. Secondary hypotheses are that this early training protocol is as feasible and as safe as standard therapy protocol. Further, The investigators expect improvements in weaning rate from mechanical ventilator, less time on mechanical ventilation, a shorter length of stay in the respiratory care center and the hospital, and a higher quality of life at 6 months after hospital discharge compared to participants receiving usual care.

Methods and design The investigators will conduct a prospective, single-center, allocation concealed and assessor-blinded randomised controlled trial with superiority design and 6-month follow-up. The study has been approved by the Ethics Committee of Taichung Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taiwan. This trial is conducted according to Taiwan law and Good Clinical Practice (GCP) guidelines.

Study population The study is being conducted in the interdisciplinary respiratory care center of Taichung Tzu Chi Hospital, Taiwan. To be eligible to participate in the study patients must be aged 18 or older, be expected to stay on mechanical ventilator for at least 21 days, which reflects a prolonged stay at mechanical ventilator. The participants with prior muscle weakness, such as a preexisting neurological or neuromuscular disease with functional deficits or a prolonged bedridden for at least 2 months prior to the respiratory care center admission, are excluded from the study. Further exclusion criteria are contraindications to cycling (mainly fractures or recent surgical procedures to the lower limbs, acute thrombosis, preexisting open wounds, extracorporeal membrane oxygenation (ECMO) and body weight of more than 150 kg), patients who are already enrolled in another intervention study, patients receiving palliative care, patients with a diagnosis on admission that excludes the possibility of walking at hospital discharge (for example, paraplegia) and lastly patients who do not understand either traditional Chinese and Taiwanese language. Standard care (control group) Participants randomised to the control group will receive usual physiotherapy and respiratory care center standard care, which includes weaning protocols and bed exercise program based on previous publications. Current physiotherapy practice consists of positioning, respiratory therapy, passive range of movement exercises for nonresponsive participants or active exercises if arousable, and early mobilization. In order to start as early as possible, physiotherapists screen participants regularly focusing on prevention and treatment of functional and pulmonary impairment. However, subject to the internal procedure, physiotherapy and mobilization will start after medical prescription. Treatments are based on the therapist's assessment and are accordingly individually tailored. Sessions will usually take place once daily from Monday to Friday and, if deemed necessary (e.g. severe weakness, intensive rehabilitation and weaning period, retained airway secretion or atelectasis in extubated participants), this includes treatment at the weekend.

Study intervention (experimental group) Participants randomised to the experimental group will receive a standardised exercise program involving early mobilization and endurance training. The clinician in charge will decide before study inclusion, whether there are any contraindications to include the patient, and during the study, if at any time the treatment should be stopped, e.g. in case of an adverse event (decreased SaO2). Therefore, the intervention will be started as soon as it is deemed safe by the treating respiratory care center team and will occur from Monday to Friday and, if deemed necessary, at the weekend. Throughout all activities, progression will be increased successively, depending on an individual's tolerance and stability. If needed, the physiotherapist will split the delivery of the exercise program into one or more sessions.

The number of treatments, its content and duration will be noted for both the control and experimental group. The endurance training will be conducted with grading exercise level. In the course of endurance training, patient's participation will be prompted verbally. After achieving patient's active participation in sitting on the bed, the goal will be to train for at least 20 min. If this is accomplished, exercise level and training period increased until a maximum of 7 on modified RPE. Tolerance and stability will be judged by the responsible physiotherapist according to patient's modified perceived level of exertion (modified RPE Scale). If a participant is able to perform the exercises correctly, he will be given a tutorial with pictures in order to train independently with nurses or family members. If unable to perform the exercises, the physiotherapist will use tactile facilitation or passive range of movement for all joints and their possible directions. If the previous exercises are well-tolerated, bed mobility and sitting upright in bed will be started. If these are well-tolerated and no contraindications as per medical prescription exist, the treatment will be further advanced to mobilizing participants to the bedside. There, balance exercises will be performed or, if needed, support will be provided by the physiotherapist or various assistive equipment. After being able to sit for at least 10 min on the side of the bed, regardless of whether support is needed, participants will be moved into a chair with an individually adapted transfer according to the individual's resources. The aim during all mobilizations will be to involve the patient as actively as possible to promote independence. While sitting, functional tasks and activities of daily living will be performed and gradually increased to standing and walking exercises.

ELIGIBILITY:
Inclusion Criteria:

* Stay on mechanical ventilation for at least 21 days
* Stable hemodynamic condition
* Can follow simple oral order

Exclusion Criteria:

* Consciousness disturbance
* Impaired cognition
* Glucose levels < 70 or >200 mg/dL
* Preexisting neurological or neuromuscular disease with functional deficits
* Contraindications to exercise (acute thrombosis, preexisting open wounds)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Weaning Rate | up to 6 weeks
  weaning from mechanical ventilator
Days of Mechanical Ventilator | up to 6 weeks
  days for mechanical ventilator using
Length of Stay | up to 6 weeks
  length of stay for RCC

SECONDARY OUTCOMES:
Physical Activity | up to 6 weeks
  physical activity (FSS-ICU)
Activity of Daily Life | up to 6 weeks
  activity of daily life (Barthel Index)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Lin, Principal Investigator — Taichung Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taichung Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taichung, Not in USA, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Zanni JM, Korupolu R, Fan E, Pradhan P, Janjua K, Palmer JB, Brower RG, Needham DM. Rehabilitation therapy and outcomes in acute respiratory failure: an observational pilot project. J Crit Care. 2010 Jun;25(2):254-62. doi: 10.1016/j.jcrc.2009.10.010. Epub 2009 Nov 26. PMID 19942399
- [Background] Jolley SE, Bunnell AE, Hough CL. ICU-Acquired Weakness. Chest. 2016 Nov;150(5):1129-1140. doi: 10.1016/j.chest.2016.03.045. Epub 2016 Apr 7. PMID 27063347
- [Result] Kayambu G, Boots R, Paratz J. Physical therapy for the critically ill in the ICU: a systematic review and meta-analysis. Crit Care Med. 2013 Jun;41(6):1543-54. doi: 10.1097/CCM.0b013e31827ca637. PMID 23528802
- [Result] Elkins M, Dentice R. Inspiratory muscle training facilitates weaning from mechanical ventilation among patients in the intensive care unit: a systematic review. J Physiother. 2015 Jul;61(3):125-34. doi: 10.1016/j.jphys.2015.05.016. Epub 2015 Jun 16. PMID 26092389
- [Result] Morris PE, Berry MJ, Files DC, Thompson JC, Hauser J, Flores L, Dhar S, Chmelo E, Lovato J, Case LD, Bakhru RN, Sarwal A, Parry SM, Campbell P, Mote A, Winkelman C, Hite RD, Nicklas B, Chatterjee A, Young MP. Standardized Rehabilitation and Hospital Length of Stay Among Patients With Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2016 Jun 28;315(24):2694-702. doi: 10.1001/jama.2016.7201. PMID 27367766
- [Result] Moss M, Nordon-Craft A, Malone D, Van Pelt D, Frankel SK, Warner ML, Kriekels W, McNulty M, Fairclough DL, Schenkman M. A Randomized Trial of an Intensive Physical Therapy Program for Patients with Acute Respiratory Failure. Am J Respir Crit Care Med. 2016 May 15;193(10):1101-10. doi: 10.1164/rccm.201505-1039OC. PMID 26651376
- [Result] Mendez-Tellez PA, Needham DM. Early physical rehabilitation in the ICU and ventilator liberation. Respir Care. 2012 Oct;57(10):1663-9. doi: 10.4187/respcare.01931. PMID 23013903